CLINICAL TRIAL: NCT05879835
Title: Safety and Effectiveness of 4% Tetrasodium Ethylenediaminetetraacetic Acid Catheter Lock Solution in Preventing Central Venous Catheter Occlusions in Children With Intestinal Failure: A Randomized Controlled Trial
Brief Title: KiteLock 4% EDTA Lock Solution for the Prevention of Occlusions in Children With Intestinal Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SterileCare Inc. (Industry)
Collaborators: Dicentra Inc. (Industry); Meditrial SrL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CT23-001-SC001
Record Dates: First submitted 2023-05-09; First posted 2023-05-30 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2024-11

CONDITIONS: Pediatric Intestinal Failure
Keywords: catheter lock solution; pediatric intestinal failure; intestinal failure; central venous catheter; KiteLock 4%; heparin; total parenteral nutrition; parenteral nutrition
MeSH Terms: conditions — Intestinal Failure; Hyperphagia

STUDY DESIGN:
Intervention Model Description: Multisite, randomized, open-label, 2-arm parallel-group superiority trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- KiteLock 4% Sterile Catheter Lock Solution (Experimental): 4% Tetrasodium EDTA lock solution (KiteLock 4% Sterile Catheter Lock Solution; SterileCare Inc., Canada) will be administered 4-24 hours daily while the patient is cycled off their PN, as per site standard operating procedures.
  Interventions: Device: KiteLock 4% Sterile Catheter Lock Solution
- Heparin Lock Solution (Active Comparator): Heparin lock solution will be administered daily per investigator judgement, given its significant clinical risk in the youngest/smallest/vulnerable subjects.
  Interventions: Device: Heparin Lock Solution

INTERVENTIONS:
Device: KiteLock 4% Sterile Catheter Lock Solution — KiteLock™ is a clear, colorless, and sterile 4% (40 mg/ml) tetrasodium EDTA solution that contains no preservatives, latex, antibiotics, or ethanol and is nonpyrogenic. Tetrasodium salt of EDTA has been shown to disrupt in vivo and ex vivo-generated biofilms by destabilizing the structural integrity of micro-organisms at the cellular level.
  Arms: KiteLock 4% Sterile Catheter Lock Solution
Device: Heparin Lock Solution — Nonpyrogenic, hypertonic preparation of heparin sodium injection, USP with sodium chloride in water for injection.
  Arms: Heparin Lock Solution

SUMMARY:
A multi-site, randomized, 2-arm open-label trial to determine if 4% Tetrasodium (EDTA) catheter lock solution is more effective than heparin lock (standard of care) in preventing central venous catheter occlusions in children with intestinal failure (IF) on total parenteral nutrition (TPN).

DETAILED DESCRIPTION:
A total of 124 (62 per arm) will be enrolled into the study. Screening and informed consent (and assent if applicable) will be obtained prior to study procedures. The baseline assessment will be completed at recruitment to the study. Once the baseline assessment is complete and eligible subjects are randomized, the study drug will be dispensed per protocol. The study follow-up period will be 52 weeks. Four follow-up clinical in-person visits will occur at 2,12, 28, 40 and 52 weeks. Visits will be conducted by physicians or nurse practitioners. The study visits will assess general status, study bloodwork, adverse events, catheter patency, alteplase use, infection assessment, catheter integrity, and provide investigational product. Telephone follow up will occur on day-3 of intervention, and once per 4 weeks, as well as in the event of outpatient care/hospital admission, or safety event. Subject daily diaries will be utilized for detailed monitoring. Diary recordings will include adverse events, including occlusive events, and any subject specific details (e.g. dwell times, heparin flushing vs. aspiration) or issues in the delivery of the study locking solutions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients managed by the intestinal rehabilitation program at one of the participating centers.
2. Diagnosis of intestinal failure defined as need for PN support for >60 days in previous 74 days for primary intestinal disease (short bowel syndrome, primary motility disorder, mucosal enteropathy).
3. Expectation of the treating physician that the patient will require PN for at least 6 months following enrollment.
4. Age less than 18 years at diagnosis but greater than 4 weeks chronological age or 40 weeks estimated gestational age, whichever is greater.
5. Stable TPN cycling (4 hours off TPN minimum per day) enabling home TPN management
6. Presence of a tunneled central venous catheter (CVC), port-a-catheter, or peripherally inserted central catheter (PICC).
7. Clinical stability for at least 4 weeks and no acute medical comorbidities.
8. A minimum dwell time of 4 consecutive hours daily.
9. Care provider willing to provide informed consent to participate in the trial and willing to comply with randomization and study protocol.

Exclusion Criteria:

1. A temporary CVC (jugular or femoral) or peripheral catheter.
2. Patients receiving long-term PN, but not due to a primary intestinal disorder (i.e., oncology patients or premature neonates on PN due to intestinal immaturity).
3. Known hypersensitivity, allergy, or reaction to EDTA.
4. Pregnancy or nursing mother.
5. Participation in another investigational device or drug trial within 30 days prior to enrollment (unless approved by the principal investigators of the trial).
6. Severe coagulopathy (platelets <50,000, or INR > 1.5).
7. Diagnosis of immunodeficiency disorder.
8. Unstable medical condition requiring hospital admission
9. Received antibiotic therapy for CLABSI within last 14 days.

Ages: 4 Weeks to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of catheter occlusions | 52 weeks
  Occlusion is defined as requiring chemical or surgical intervention to restore patency. Occlusion rates will be pooled for each study arm and reported per 1000 catheter days.

SECONDARY OUTCOMES:
Incidence of Central Line-Associated Blood Stream Infections (CLABSI) | 52 weeks
  CLABSI is defined per the Centers for Disease Control-National Healthcare Safety Network (CDC-NSHN) definition. CLABSI rates will be pooled for each study arm and reported per 1000 catheter days.
Incidence of breakage, removal, or reinsertion of catheter | 52 weeks
  Breakage of the catheter line, surgical removal of the line or reinsertion of the line into the vein will be recorded. Event rates will be pooled for each study arm and reported per 1000 catheter days.
Incidence of central venous thrombosis | 52 weeks
  Central venous thrombosis shall be clinically diagnosed by investigators, including the collection of brain imaging. Central Venous Thrombosis rates will be pooled for each study arm and reported per 1000 catheter days.
Proportion of subjects with development of Intestinal failure-associated liver disease (IFALD) | 52 weeks
  IFALD is defined as (cholestasis defined as conjugated bilirubin >2mg/dL, advanced IFALD defined as conjugated bilirubin >6mg/dL) sustained for >2 weeks in absence of sepsis. Proportion shall be reported for each study arm
Incidence of lock-related Serious Adverse Events (SAEs) | 52 weeks
  SAEs are defined per Good Clinical Practice. SAE rates will be pooled for each study arm and reported per 1000 catheter days.

OTHER OUTCOMES:
Proportion of subjects requiring hospital admission related to catheter complications | 52 weeks
  Proportion shall be reported for each study arm.
Length of stay for hospitalization related to catheter complications | 52 weeks
  Length of hospital stay shall be reported in days. Mean shall be reported for each study arm

CONTACTS AND LOCATIONS:
Overall Officials: Paul Wales, MD, Principal Investigator — Cincinnati Children's
Locations (8):
- United States (8):
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Columbia University Irving Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Cook Children's Health Care System, Fort Worth, Texas
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Background] Quirt J, Belza C, Pai N, Clause RF, Markovic F, Wong-Sterling S, Avitzur Y, Wales PW. Reduction of Central Line-Associated Bloodstream Infections and Line Occlusions in Pediatric Intestinal Failure Patients Receiving Long-Term Parenteral Nutrition Using an Alternative Locking Solution, 4% Tetrasodium Ethylenediaminetetraacetic Acid. JPEN J Parenter Enteral Nutr. 2021 Aug;45(6):1286-1292. doi: 10.1002/jpen.1989. Epub 2020 Aug 30. PMID 32770561